CLINICAL TRIAL: NCT06616584
Title: A Randomized Phase II/III Study of Docetaxel and Ramucirumab With or Without Cemiplimab for Participants Previously Treated With Platinum-Based Chemotherapy and Immunotherapy for Stage IV or Recurrent Non-Small Cell Lung Cancer (Lung-MAP Non-Matched Sub-Study)
Brief Title: Adding the Immunotherapy Drug Cemiplimab to Usual Treatment for People With Advanced Non-Small Cell Lung Cancer Who Had Previous Treatment With Platinum Chemotherapy and Immunotherapy (An Expanded Lung-MAP Treatment Trial)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: Regeneron Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1800E; NCI-2024-06444 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1800E (Other: SWOG); S1800E (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2024-08-27; First posted 2024-09-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; cemiplimab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Docetaxel; Magnetic Resonance Spectroscopy; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ramucirumab, docetaxel) (Active Comparator): Patients receive dexamethasone PO BID on days 0-2, ramucirumab IV over 30-60 minutes on day 1 and docetaxel IV over 60 minutes on day 1 of each cycle (each cycle is 21 days). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dexamethasone; Drug: Docetaxel; Procedure: Magnetic Resonance Imaging; Biological: Ramucirumab
- Arm II (cemiplimab, ramucirumab, docetaxel) (Experimental): Patients receive dexamethasone PO BID on days 0-2, ramucirumab IV over 30-60 minutes on day 1, docetaxel IV over 60 minutes on day 1, and cemiplimab IV over 30 minutes on day 1 of each cycle (each cycle is 21 days). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Drug: Dexamethasone; Drug: Docetaxel; Procedure: Magnetic Resonance Imaging; Biological: Ramucirumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
  Arms: Arm II (cemiplimab, ramucirumab, docetaxel)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC 1121B; IMC-1121B; IMC1121B; LY 3009806; LY-3009806; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase II/III Expanded Lung-MAP treatment trial compares the effect of adding cemiplimab to docetaxel and ramucirumab versus docetaxel and ramucirumab alone in treating patients with non-small cell lung cancer that is stage IV or that has come back after a period of improvement (recurrent). Cemiplimab is a monoclonal antibody that stimulates the immune system by blocking the PD-1 pathway. Tumors use the PD-1 pathway to escape attacks from the immune system. By blocking the PD-1 pathway, cemiplimab may help the immune system recognize and attack tumor cells. Docetaxel is in a class of medications called taxanes. It stops tumor cells from growing and dividing and may kill them. Ramucirumab is a monoclonal antibody that may prevent the growth of new blood vessels that tumors need to grow. Adding cemiplimab to usual treatment, docetaxel and ramucirumab, may kill more tumor cells compared to docetaxel and ramucirumab alone in treating patients with stage IV or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival (OS) between participants randomized to docetaxel and ramucirumab with or without cemiplimab (REGN2810) who have acquired resistance to platinum-based chemotherapy and immunotherapy for stage IV or recurrent non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To compare investigator-assessed progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 between the arms.

II. To compare investigator-assessed response rates (confirmed or unconfirmed, complete response [CR] or partial response [PR]) per RECIST 1.1 between the arms among participants with measurable disease.

III. To compare the investigator-assessed disease control rate (confirmed or unconfirmed, complete response [CR], or partial response [PR], and stable disease) between the arms.

IV. To evaluate the duration of response (DoR) among responders within each arm.

V. To evaluate the frequency and severity of toxicities within each arm. VI. To compare investigator-assessed PFS between the arms within the subgroups defined by the stratification factors (histology and performance status) and by PD-L1 subgroups defined as PD-L1 negative (< 1% tumor proportion score [TPS]), intermediate PD-L1 (1-49% TPS), and PD-L1 high (>= 50% TPS).

VII. To compare OS between the arms within the subgroups defined by the stratification factors (histology and performance status) and by PD-L1 subgroups defined as PD-L1 negative (< 1% TPS), intermediate PD-L1 (1-49% TPS), and PD-L1 high (>= 50% TPS).

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To collect, process, and bank cell-free deoxyribonucleic acid (cfDNA) at baseline, cycle 3 day 1, and progression for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor DNA (ctDNA).

II. To establish a tissue/blood repository to pursue future studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive dexamethasone orally (PO) twice daily (BID) on days 0-2, ramucirumab intravenously (IV) over 30-60 minutes on day 1 and docetaxel IV over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

ARM II: Patients receive dexamethasone PO BID on days 0-2, ramucirumab IV over 30-60 minutes on day 1, docetaxel IV over 60 minutes on day 1, and cemiplimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, and CT or MRI throughout the study.

After completion of study treatment, patients are followed up every 3-6 months for up to 3 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been assigned to S1800E by the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC). Assignment to S1800E is determined by the LUNGMAP protocol
* Participants must have measurable or non-measurable disease documented by CT or MRI. The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to randomization. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to randomization. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration
* Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to randomization
* Participants must have received exactly one anti-PD-1 or anti-PD-L1 therapy for advanced disease (stage IV or recurrent disease, or stage I-III disease in certain circumstances outlined below). Anti-PD-1 or anti-PD-L1 therapy may have been given alone or in combination with other therapy. For participants who received neoadjuvant, adjuvant, and/or consolidation anti-PD-1 or anti-PD-L1 therapy for stage I-III disease:

  * If they experienced disease progression within (≤) 365 days from initiation (cycle 1 day 1) or anti-PD-1 or anti-PD-L1 therapy, this counts as the single allowed anti-PD-1 or anti-PD-L1 therapy for advanced disease
  * If they experienced disease progression more than (>) 365 days from initiation (cycle 1 day 1) or anti-PD-1 or anti-PD-L1 therapy, this is not considered anti-PD-1 or anti-PD-L1 therapy for advance disease. These participants must have received anti-PD-1 or anti-PD-L1 therapy for stage IV or recurrent disease
* Participants must have experienced disease progression (in the opinion of the treating investigator) more than (>) 84 days following initiation (cycle 1 day 1) of their most recent anti-PD-1 or anti-PD-L1 therapy
* Participants who received anti-PD-1 or anti-PD-L1 therapy for stage IV or recurrent disease must have had a best response of stable disease, partial response or complete response (in the opinion of the treating investigator) on the anti-PD-1 or anti-PD-L1 therapy for stage IV or recurrent disease
* Participants must have received platinum-based chemotherapy and experienced disease progression (in the opinion of the treating investigator) during or after this regimen
* Participants with a known sensitizing molecular alteration for which a Food and Drug Administration (FDA)-approved targeted therapy for NSCLC exists (e.g., EGFR, ALK, ROS1, BRAF, RET, NTRK, KRAS, HER2, and MET sensitizing mutations), must have previously received at least one of the approved therapy(s). Prior targeted therapy for participants with targetable alterations is allowed if all other eligibility criteria are also met
* Participants must have recovered (≤ grade 1) from any side effects from the most recent anti-cancer treatment prior to randomization
* Participants must not have received prior therapy with docetaxel for this disease
* Participants must not have received any palliative radiation therapy within 14 days (or palliative bone radiation therapy within 7 days) prior to randomization
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, or biologic therapy for cancer treatment while receiving treatment on this study
* Participants must not have undergone major surgery within 28 days prior to randomization, or subcutaneous venous access device placement within 7 days prior to randomization. Participants must not have postoperative bleeding complications or wound complications from a surgical procedure performed within 2 months prior to randomization. The participant must not have elective or planned major surgery to be performed during the course of this study
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to randomization)
* Hemoglobin ≥ 9.0 g/dL (within 28 days prior to randomization)
* Platelets ≥ 100 x 10^3/uL (within 28 days prior to randomization)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to randomization) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional ULN (within 28 days prior to randomization). Participants with history of liver metastasis must have AST and ALT ≤ 5 x ULN
* Participants must have a creatinine ≤ the institutional (I)ULN or calculated creatinine clearance ≥ 50 mL/min using the following Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to randomization
* Participants must have a urinary protein test performed within 28 days prior to randomization
* Participants' most recent Zubrod/Eastern Cooperative Oncology Group (ECOG) performance status must be 0-1 and be documented within 28 days prior to randomization
* Participants must have a completed medical history and physical exam within 28 days prior to randomization
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to randomization, if indicated by the treating investigator
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to randomization, if indicated by the treating investigator
* Participants with known human immunodeficiency virus (HIV) infection are eligible, provided they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to randomization
* Participants must not have a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have an active autoimmune disease that has required systemic treatment within 730 days prior to randomization (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Participants must not have any history of primary immunodeficiency
* Participants must be able to safely receive study therapy and must not have experienced the following:

  * Any grade 3 or worse immune-mediated adverse event. Exception: asymptomatic nonbullous/nonexfoliative rash
  * Any unresolved grade 2 immune-mediated adverse event
  * Any toxicity that led to permanent discontinuation of prior anti-PD-1/PD-L1 immunotherapy
  * Exception to the above: Toxicities of any grade that requires replacement therapy and has stabilized on therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are allowed
* Participants must not have any history of organ transplant that requires use of immunosuppressives
* Participants must not have received a live or live attenuated vaccine within 28 days prior to randomization. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever rabies, Bacillus Calmette-Guerin (BCG) and typhoid vaccine. Seasonal influenza vaccines and COVID-19 vaccines are allowed, however, intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated and are not allowed
* Participants must not have clinical signs or symptoms of active tuberculosis infection
* Participants must not have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis/interstitial lung disease
* Participants must not have had a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to randomization
* Participants must not have a history of gastrointestinal perforation or fistula within 6 months prior to randomization
* Participants must not have grade 3-4 gastrointestinal bleeding (defined by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]5) within 3 months prior to randomization. No history of gastrointestinal (GI) bleed within 3 months prior to randomization
* Participants must not have any grade III/IV cardiac disease as defined by the New York Heart Association criteria (i.e., participants with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months prior to randomization, or serious uncontrolled cardiac arrhythmia
* Participants must not have experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to randomization
* Participants must not have gross hemoptysis within two months prior to randomization (defined as bright red blood or ≥ 1/2 teaspoon) or with radiographic evidence of intratumor cavitation or has radiologically documented evidence of major blood vessel invasion or encasement by cancer
* Participants must not have been diagnosed with venous thrombosis within 3 months prior to randomization. Participants with venous thrombosis diagnosed more than 3 months prior to randomization must be on stable doses of anticoagulants
* Participants must not have cirrhosis at a level of Child-Pugh B (or worse) AND a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis, OR any degree of cirrhosis
* Participants must not be pregnant or breastfeeding (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Participants must be offered participation in specimen banking. With participant consent, specimens must be collected and submitted via the SWOG specimen tracking system
* NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. NOTE: Participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 3 years
  OS will be compared between arms and within the subgroups defined by the stratification factors and by PD-L1 subgroups. Distributions of OS will be estimated using the method of Kaplan-Meier. Hazard ratios for comparisons of OS will be estimated using a Cox Proportional Hazards regression model, with baseline hazard stratification using the stratification factors. Testing will be done using a stratified log-rank test. Confidence intervals (CIs) about medians will be estimated using the method of Brookmeyer-Crowley. For point estimates at landmark times, the associated CIs will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization to date of first documentation of progression, symptomatic deterioration, or death, whichever comes first, assessed up to 3 years
  PFS will be compared between arms and within the subgroups defined by the stratification factors and by PD-L1 subgroups. PFS between the arms will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Distributions of PFS will be estimated using the method of Kaplan-Meier. Hazard ratios for comparisons of PFS will be estimated using a Cox Proportional Hazards regression model, with baseline hazard stratification using the stratification factors. Testing will be done using a stratified log-rank test. CIs about medians will be estimated using the method of Brookmeyer-Crowley. For point estimates at landmark times, the associated CIs will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function.
Response rates | Up to 3 years
  Response rates (complete response [CR] or partial response [PR]) between the arms will be assessed per RECIST 1.1. Binary proportions along with confidence intervals will be estimated for response. CIs will be estimated using the Wilson Score method with continuity correction.
Disease control rates | Up to 3 years
  Disease control rates (CR or PR and stable disease) between the arms. Binary proportions along with confidence intervals will be estimated for disease control rate. CIs will be estimated using the Wilson Score method with continuity correction.
Duration of response (DOR) | From date of first documentation of response by RECIST 1.1 (CR or PR, confirmed or unconfirmed) to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will be assessed among participants who achieve a response. Distributions of DOR will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 90 days after last dose of study treatment
  Adverse events will be assessed and graded using Common Terminology Criteria for Adverse Events version 5.0. Individual toxicities within each treatment arm will be summarized by grade, among those reported as being attributable to treatment (possibly, probably, or definitely attributable to treatment). The frequency and severity for each adverse event term will be summarized for grade 3, 4 and 5 separately, and as worst grade reported overall all reported adverse events.

OTHER OUTCOMES:
Cell-free deoxyribonucleic acid | At baseline, cycle 3 day 1 and at progression up to 3 years (each cycle is 21 days)
Tissue/blood repository | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Saiama N Waqar, Principal Investigator — SWOG Cancer Research Network
Locations (361):
- United States (361):
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Malbis, Daphne, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Saraland, Saraland, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Enloe Medical Center, Chico, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mather Veteran Affairs Medical Center, Mather, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Malcom Randall Veterans Administration Medical Center, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Saint Agnes Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Durham VA Medical Center, Durham, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - United Hospital Center, Bridgeport, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin